CLINICAL TRIAL: NCT07092423
Title: The Effect of Semi-elemental Enteral Nutrition on Gastrointestinal Tolerance in Patients With Traumatic Brain Injury: a Randomized Exploratory Study
Brief Title: Effect of Semi-elemental Enteral Nutrition on Gastrointestinal Tolerance in Patients With Traumatic Brain Injury.
Acronym: SEMINAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SEMINAR Study
Record Dates: First submitted 2025-04-11; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury; Neurocritical Care; Enteral Feeding Intolerance
Keywords: Traumatic Brain Injury; Enteral Nutrition; Gastrointestinal Intolerance; Semi-elemental Formula; Neurocritical Care; Prognosis
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Patients will receive semi-elemental enteral nutrition.
  Interventions: Dietary Supplement: Semi-elemental formula
- Control Group (Active Comparator): Patients will receive standard enteral nutrition.
  Interventions: Dietary Supplement: Standard formula

INTERVENTIONS:
Dietary Supplement: Semi-elemental formula — Treatment: Semi-elemental enteral nutrition Objective: To assess the efficacy of semi-elemental enteral nutrition in enhancing gastrointestinal tolerance in patients with severe traumatic brain injury.
  Arms: Intervention Group
Dietary Supplement: Standard formula — Treatment: Standard enteral nutrition Objective: To serve as the control for evaluating the efficacy and safety of semi-elemental enteral nutrition versus standard nutritional therapy
  Arms: Control Group

SUMMARY:
Study Objective This clinical trial primarily aims to investigate whether semi-elemental enteral nutrition (SEN) improves gastrointestinal tolerance in patients with severe traumatic brain injury (TBI) and to evaluate its impact on clinical outcomes. The safety profile of SEN will also be assessed.

Key Research Questions Does SEN reduce the incidence of acute gastrointestinal injury (AGI) in severe TBI patients?

Study Design

Participants will be randomized 1:1 into either:

Intervention group: Receives SEN initiated within 48 hours post-injury and continued for ≥7 days.

Control group: Receives standard enteral nutrition over the same period.

DETAILED DESCRIPTION:
Background:

Patients with traumatic brain injury (TBI) frequently exhibit gastrointestinal dysfunction secondary to central nervous system impairment. This dysregulation impairs nutrient absorption, exacerbates systemic inflammation, and compromises clinical recovery trajectories. Emerging evidence suggests that semi-elemental enteral nutrition (SEN)-featuring hydrolyzed macronutrients with low-osmolality formulations-may mitigate these sequelae by reducing digestive burden and enhancing mucosal healing. However, robust clinical evidence supporting its superiority over standard enteral feeding in severe TBI populations remains limited.

Objectives:

Primary Objective:

To evaluate the efficacy of semi-elemental enteral nutrition (SEN) in improving gastrointestinal tolerance during the acute phase (first 7 days post-injury) in patients with severe traumatic brain injury (TBI).

Secondary Objectives:

1. To assess gastrointestinal complications within 7 days of enteral nutrition initiation, including:

   Incidence of diarrhea and diarrhea-free days Incidence of constipation Incidence of vomiting Incidence of gastroparesis Incidence of abdominal distension Time to first onset of gastrointestinal intolerance symptoms Duration of gastrointestinal intolerance symptoms
2. To evaluate clinical outcomes:

   Hospitalization duration (total and ICU-specific) 6-month mortality and functional recovery
3. To determine safety profiles:

Infection rates Pneumonia incidence Other adverse events

Study Design:

A multicenter, randomized, double-blind, parallel-group exploratery trial will be conducted. 100 severe TBI patients will be allocated 1:1 to intervention (SEN formula) or control (standard formula) arms within 48 hours of injury.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* Clinically diagnosed with closed traumatic brain injury;
* Glasgow Coma Scale (GCS) score ≤ 8;
* Ability to initiate enteral nutrition within 48 hours post-injury;
* Expected need for enteral nutrition support ≥3 days based on clinical assessment (Nutritional Risk Screening 2002 [NRS2002] score ≥3).

Exclusion Criteria:

* GCS=3 with bilateral fixed and dilated pupils;
* Hemodynamic instability or respiratory failure: mean arterial pressure <70mmHg, PaO2/FiO2<150, PaCO2<30 mmHg or >45 mmHg, or lactate >5 mmol/l;
* Contraindications to both nasogastric and nasojejunal tube placement, or inability to complete tube placement within 48 hours of onset;
* Contraindications to enteral nutrition therapy or semi-recumbent positioning;
* Pre-existing intellectual disability or physical disability affecting outcome assessment;
* Gastrointestinal abnormalities likely to affect gastrointestinal function, such as short bowel syndrome (defined as total small bowel length ≤122 cm), ulcerative colitis, Crohn's disease, or any form of ostomy;
* Body mass index (BMI) <18kg/m2;
* Concomitant abdominal injury or extracranial injury with AIS score >3 in any region;
* Presence of malignancy, severe cardiac insufficiency (ejection fraction <50%), severe hepatic failure (Child-Pugh score ≥7), or severe renal failure (glomerular filtration rate ≤30 mL/min or serum creatinine ≥4mg/dL) at NICU admission;
* Concurrent severe disease with expected survival ≤14 days;
* Pregnancy, within 30 days postpartum, or breastfeeding;
* Refusal of treatment or receipt of palliative care;
* Patient or family declines informed consent;
* Current participation in another interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Gastrointestinal Intolerance | Within 7 days.
  Proportion of patients developing gastrointestinal intolerance within 7 days of enteral nutrition initiation.
  (Composite endpoint including: vomiting, diarrhea, constipation, gastroparesis, gastrointestinal bleeding, and abdominal distension.)

SECONDARY OUTCOMES:
Hospitalization length of stay (LOS) | Periprocedural.
  Total length of stay in the hospital.
NICU LOS | Periprocedural
  Total length of stay in the neurological intensive care unit (NICU)
In-hospital mortality | Periprocedural.
  Mortality rate in hospital.
ICU mortality | Periprocedural
  Mortality rate in NICU
Three-month mortality | Within 3 months.
  Mortality rate at 3-month.
Six-month mortality | Within 6 months.
  Mortality rate at 6-month.
Functional outcomes (GOSE) | Within 6 months.
  The Glasgow Outcome Scale-Extended (GOSE) scores at 3 and 6 months. The score ranges from 1 to 8, with higher scores indicating a better outcome.
Functional outcomes (Barthel) | Within 6 months.
  The Barthel Index scores at 3 and 6 months.The score ranges from 1 to 100, with higher scores indicating a better outcome.
Gastrointestinal intolerance events | Within 7 days.
  Gastrointestinal intolerance events within 7 days of enteral nutrition initiation, including:
  1. Incidence of diarrhea.
  2. Diarrhea-free days.
  3. Incidence of constipation.
  4. Incidence of vomiting.
  5. Incidence of gastroparesis.
  6. Incidence of abdominal distension.
  7. Time to first onset of symptoms.
  8. Symptom duration.
Infection | Within 14 days
  Infection rate during 14-day period (or throughout hospitalization if discharged earlier).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, MD, PhD, Study Chair — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Will be determined in accordance with sponsor requirements.